CLINICAL TRIAL: NCT05853315
Title: Long-term Results After Surgical Basal Cell Carcinoma Excision in the Eyelid Region: Revisited
Brief Title: BCC Excision Revisited
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Reinhard Told, Priv. Doz. Dr., Medical University of Vienna
Other Study IDs: 1997/2019
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Basal Cell Carcinoma; Eye Diseases; Eye Cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Eye Diseases; Eye Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery — Surgical Excision

SUMMARY:
To readdress basal cell carcinoma (BCC) in the periocular region to prove histologically controlled surgical treatment efficacy and to identify high-risk characteristics.

ELIGIBILITY:
Inclusion criteria:

* Patient records were reviewed for the presence of BCC and surgical excision with frozen sections control of the wound margins in the periocular region,
* conducted between 01.01.2009 and 31.12.2019.
* Periocular was defined as the area involving the medial and lateral canthus as well as the upper and lower eyelids.

Exclusion criteria:

* BCCs outside of this region were excluded from this analysis,
* as well as incomplete records.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: male and female patients with periocular basal cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
BCC Recurrence | mean 3-5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria